CLINICAL TRIAL: NCT03332628
Title: Evaluating Racial and Ethnic Differences in Micropore Closure Rates After Microneedle Application to the Skin
Brief Title: Racial/Ethnic Differences in Microneedle Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Nicole K Brogden, Associate Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201708721
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: Peer Reviewed Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microneedle application (Other): This is the only study arm, which all participants complete. Nine sites on the upper arm will be identified. Baseline measurements of transepidermal water loss, electrical resistance, hydration, and color will be made at each site. The 9 sites will be divided into clusters of 3 sites each. The first cluster will have small microneedle patches applied to at each site. This will only occur on the first study day. Transepidermal water loss and electrical resistance are re-measured immediately after microneedle application. The sites will be covered with a small patch secured with medical tape. The second cluster of sites will not receive microneedle application but will just be covered with patches. The last cluster of sites will not have microneedle application or patches. Electrical resistance will be re-measured at all sites for 4 days after microneedle application. Measurements from the 2nd and 3rd cluster of sites allow each subject to serve as their own control in data analysis.
  Interventions: Device: Microneedle patch

INTERVENTIONS:
Device: Microneedle patch — Each patch contains 50 microneedles.

SUMMARY:
The study to be performed will define the rate of skin barrier recovery following microneedle treatment of the skin in healthy subjects of differing racial/ethnic backgrounds.

DETAILED DESCRIPTION:
Transdermal drug delivery (by way of patches that adhere to the skin and deliver drug in a time-dependent fashion) allows for systemic drug delivery through the skin, while avoiding many of the side effects and challenges associated with oral or intravenous drug delivery. One significant challenge limiting the number of drug compounds that can be transdermally delivered is the hydrophobic nature of the skin, which provides a highly efficient barrier against the absorption of drug molecules. Microneedles are a minimally invasive means of allowing drug molecules to cross the skin by creating micron-sized channels (also called micropores) in the skin, thereby increasing its permeability. Microneedles have been safely used in hundreds of patients for administration of drugs and vaccines through the skin. Studies have demonstrated that microneedle treatment is relatively painless and well-tolerated by most patients.

Following microneedle treatment, the skin must heal the micropores in order to restore barrier function. In young healthy individuals this process takes approximately 48 to 72 hours when the skin is covered by an occlusive patch. The timeframe for micropore closure is longer in elderly individuals (>65 years of age), taking several days longer to restore the skin barrier. As evidenced by the differences in micropore closure rate observed with advancing age, biological variation can have a significant effect on the skin's healing properties. There are almost no data available regarding how race and ethnicity affect skin response to microneedle insertion. It is crucial to better understand how the rates of micropore closure vary in different racial/ethnic populations because the potential for variability in drug delivery is high if the recovery timeframes are poorly understood.

In this study we will measure hydration and color to characterize the epidermal properties of individuals of different self-identified race and ethnicity. Measurements of trans-epidermal water loss and electrical impedance will be used to evaluate the formation of micropores in the skin; the electrical impedance measurements will be used to calculate the rate of micropore closure. All of these skin characteristics can be measured using noninvasive methods that are quick and painless.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be healthy men and women between 18 - 50 years of age who identify as African American or Black, Asian, Hispanic or Latino, American Indian/Alaska Native, Native Hawaiian/Other Pacific Islander, Caucasian/White, bi-/multiracial.

Exclusion Criteria:

* Unable to give consent
* Severe general allergies requiring chronic treatment with steroids or antihistamines
* Previous adverse reaction to microneedle insertion
* Known allergy or adverse reaction to medical tape, adhesive, or aloe vera
* Anyone with inflammatory diseases of the skin or diseases that alter immune function
* Anyone taking any medications that impair the immune system will be excluded (contraceptives, vitamins, and topical products on the face will be allowed)
* Anyone with current malignancy or history of malignancy present at the treatment site (upper arm)
* Anyone with any of the following present at the treatment site (upper arm): eczema or scaling, inflammation, erythema, edema, blisters
* Anyone with uncontrolled mental illness that would, in the opinion of the physician, affect their ability to understand or reliably participate in the study
* Anyone taking medications in the following therapeutic classes will be excluded: HMGCoA reductase inhibitors ("statins"), oral or topical steroids, oral antibiotics, topical antibiotics at the local treatment site, topical antihistamines at the local treatment site, beta-blockers, and systemic or topical NSAIDS/analgesics
* Anyone who is pregnant or nursing
* Anyone with any condition that would, in the opinion of the PI or physician, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole K Brogden, PharmD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment on this study was open from January 2018 to November 2019. Study procedures were conducted at the University of Iowa Hospitals and Clinics in the Clinical Research Clinic by members of the research staff.
Pre-assignment Details: Subjects were screened after consenting to participate in the study. Participants that did not meet screening criteria were withdrawn from the study, 5 of our 132 consented participants fell into this exclusionary criteria. 9 of 132 participants signed the consent and stopped returning communication with study staff prior to scheduling their appointments, they were withdrawn from the study due to lack of follow-up. 5 of 132 voluntarily withdrew consent because of schedule conflicts.
Groups:
- Microneedle Application: This is the only arm of the study, which all participants complete. In each subject, 9 sites on the upper arm will be identified. Baseline measurements of transepidermal water loss, electrical resistance, hydration, and color will be made at each site. The 9 sites will be divided into 3 clusters of 3 sites each. The first cluster will have small microneedle patches applied to at each site. This will only occur on the first study day, and the microneedle patches will then be discarded. The sites will be covered with a small patch secured with medical tape. The second cluster of sites will not receive microneedle application but will just be covered with patches. The last cluster of sites will not have microneedle application or patches. Electrical resistance will be re-measured daily at all sites for 4 consecutive days after microneedle application. The measurements from the second and third cluster of sites allow each subject to serve as their own control in data analysis.
  Microneedle patch: Each patch contains 50 microneedles.
Period: Overall Study
Arm/Group | Microneedle Application
Started | 113
Completed | 111
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Microneedle Application
Number analyzed (Participants) | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 111
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.9 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 32
  Bi-/Multi-racial | 10
  Black | 22
  White | 23
  Latino | 23
  Native American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 111

OUTCOME MEASURES:

1. Primary Outcome: Micropore Closure Time
Description: The time required for the skin barrier to be restored after microneedle application will be determined using electrical resistance measurements. Differences in the skin electrical resistance will be determined through measurements made every day with skin electrodes attached to an impedance meter. These data for micropore closure are only collected from the microneedle sites. Using the data collected from all 5 days an average micropore closure time will be calculated, which can be compared between subsets of participants based on race/ethnicity.
Time Frame: Five days
Population: Data from all 111 participants was analyzed. The number in each row differs from the overall number because results are reported according to racial and ethnic subgroups.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Microneedle Application: This is the only arm of the study, which all participants complete. In each subject, 9 sites on the upper arm will be identified. The 9 sites will be divided into 3 clusters of 3 sites each. Baseline measurements of hydration and color will be made at each site. The first site cluster will have small microneedle patches applied to at each site. This will only occur on the first study day, and the microneedle patches will then be discarded. Measurements of transepidermal water loss and impedance will be made before and after the microneedle treatments at these 3 sites. The sites will be covered with a small patch secured with medical tape. The second cluster of sites will not receive microneedle application but will just be covered with patches. The last cluster of sites will not have microneedle application or patches. Electrical resistance will be measured daily for 4 consecutive days after microneedle application. Measurements from the second and third cluster of sites allow each subject to serve as their own control in data analysis.
  Microneedle patch: Each patch contains 50 microneedles.
Arm/Group | Microneedle Application
Number analyzed (Participants) | 111
hours
  Asian: number analyzed (Participants) | 32
  Asian | 44.1 (14.0)
  Bi-/Multi-racial: number analyzed (Participants) | 10
  Bi-/Multi-racial | 48.0 (16.0)
  Black: number analyzed (Participants) | 22
  Black | 66.5 (19.5)
  White: number analyzed (Participants) | 23
  White | 50.1 (12.4)
  Latino: number analyzed (Participants) | 23
  Latino | 61.1 (16.1)
  Native American/Hawaiian: number analyzed (Participants) | 1
  Native American/Hawaiian | 72 (0)

2. Secondary Outcome: Change in Trans-epidermal Water Loss
Description: Percent change from baseline trans-epidermal water loss will be calculated after microneedle application, and these data are only collected from the microneedle sites. Percent change is calculated as (trans-epidermal water loss after microneedle application/baseline trans-epidermal water loss) x 100.
Time Frame: Baseline (Day 0) and post microneedle application (Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percantage change
Arm/Group | Microneedle Application
Number analyzed (Participants) | 111
Percantage change
  Asians: number analyzed (Participants) | 32
  Asians | 212.81 (58.83)
  Bi-/Multi-racial: number analyzed (Participants) | 10
  Bi-/Multi-racial | 203.12 (79.81)
  Black: number analyzed (Participants) | 22
  Black | 240.95 (97.47)
  White: number analyzed (Participants) | 23
  White | 228.25 (75.58)
  Latino: number analyzed (Participants) | 23
  Latino | 223.93 (82.31)
  Native American/Hawaiian: number analyzed (Participants) | 1
  Native American/Hawaiian | 200 (0)

3. Secondary Outcome: Skin Color
Description: Lightness/darkness of the skin is measured with a tristimulus colorimeter and reported in a unitless value called L*. Higher L* values denote lighter skin, while lower L* values denote darker skin. Data are calculated as the mean of measurements from all 9 sites on the arm.
Time Frame: Baseline (Day 0)
Population: Data from all 111 participants was analyzed. Data are calculated as the mean of measurements from all 9 sites on the arm. The number in each row differs from the overall number because results are reported according to racial and ethnic subgroups. Results are presented as prespecified in the protocol to collect and analyze data for all subjects together by ethnicity/race.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Microneedle Application
Number analyzed (Participants) | 111
Unitless
  Black: number analyzed (Participants) | 22
  Black | 40.61 (6.74)
  Asian: number analyzed (Participants) | 32
  Asian | 59.77 (7.62)
  Bi-/Multi-racial: number analyzed (Participants) | 10
  Bi-/Multi-racial | 61.12 (5.79)
  White: number analyzed (Participants) | 23
  White | 64.67 (4.71)
  Latino: number analyzed (Participants) | 23
  Latino | 58.84 (7.21)
  Native American/Hawaiian: number analyzed (Participants) | 1
  Native American/Hawaiian | 60.37 (0)

4. Secondary Outcome: Hydration
Description: Baseline skin hydration will be measured using a capacitance probe. The software calculates arbitrary unitless values. Values less than 30 are considered very dry while values over 40 are considered sufficiently moisturized. Data are calculated as the mean of measurements from all 9 sites on the arm.
Time Frame: Baseline (Day 0)
Population: Data from all 111 participants was analyzed. The number in each row differs from the overall number because results are reported according to racial and ethnic subgroups. Data are calculated as the mean of measurements from all 9 sites on the arm. Results are presented as prespecified in the protocol to collect and analyze data for all subjects together by ethnicity/race.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Microneedle Application
Number analyzed (Participants) | 111
Unitless
  Asians: number analyzed (Participants) | 32
  Asians | 38.32 (23.97)
  Bi-/Multi-racial: number analyzed (Participants) | 10
  Bi-/Multi-racial | 50.27 (21.60)
  Black: number analyzed (Participants) | 22
  Black | 34.75 (18.49)
  White: number analyzed (Participants) | 23
  White | 36.06 (18.81)
  Latino: number analyzed (Participants) | 23
  Latino | 35.61 (14.23)
  Native American/Hawaiian: number analyzed (Participants) | 1
  Native American/Hawaiian | 24.1 (0)

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored during the 5 days while a subject was completing the study and for three days after study completion.
Description: Through the course of this study adverse events were recorded as reported from the subjects.
Arm/Group | Microneedle Application
All-Cause Mortality (participants affected / at risk) | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 1/113
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Microneedle Application (N=113)
Mild Skin reaction to waterproof tape (Skin and subcutaneous tissue disorders) | 1 — One subject discontinued the study early due to a mild skin reaction to the waterproof medical tape used to secure the occlusive patches on the skin (this subject's data was not included in the analysis)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT03332628/Prot_SAP_000.pdf